CLINICAL TRIAL: NCT03295604
Title: A Novel Volumetric Analysis Using CAD/CAM Scanners in Gingival Recession
Brief Title: A Novel Volumetric Analysis Using CAD/CAM Scanners in Gingival Recession Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacer Sahin Aydinyurt (Other)
Collaborators: Yuzuncu Yil University (Other)
Responsible Party: Sponsor-Investigator, Hacer Sahin Aydinyurt, assistant professor, Yuzuncu Yil University
Organization: Yuzuncu Yil University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YuzuncuYıl 3
Record Dates: First submitted 2017-08-16; First posted 2017-09-28 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Gingival Recession
Keywords: Gingival recession; Subepithelial connective tissue grafts; CAD/CAM
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): Miller class I-II gingival recession defects operated with sub epithelial connective tissue graft (SCTG) in addition with enamel matrix derivatives (EMD) (Emdogain ®, Switzerland ) in SCTG+EMD group.
  Interventions: Procedure: SCTG+EMD
- control group (Experimental): Miller class I-II gingival recession defects operated with only sub epithelial connective tissue graft (SCTG). No drug or something else were used
  Interventions: Procedure: SCTG

INTERVENTIONS:
Procedure: SCTG+EMD — Miller class I-II gingival recession defects were operated with SCTG+EMD
  Arms: test group
Procedure: SCTG — Miller class I-II gingival recession defects were operated with SCTG only and
  Arms: control group

SUMMARY:
Aim: In this ramdomised clinical trial (RCT), the aim was to compare clinical periodontal data of subepithelial connective tissue graft (SCTG) group and SCGT+enamel matrix derivatives (EMD) group in terms of gained gingiva volume (GGV) and gained gingiva surface area (GGSA) by scanners of computer-aided design/computer-aided manufacturing (CAD/CAM) devices.

Materials and Methods: A total of 35 Miller class I-II gingival recession defects were involved in this study (n=17 in SCTG group, n=18 in SCTG+EMD group). In addition to periodontal clinical parameters, three dimensional (3D) images were recorded using CAD/CAM system before the treatment, at the 1st month and at the 6th months after the treatment. The images were superimposed using softwares and GGV, GGSA were calculated.

DETAILED DESCRIPTION:
Study populations:

In this study, totally 35 gingival recession (GR) defects in 35 patients, who applied with complaints of poor aesthetic and/or root surface sensitivity. Following patients were admitted to the study: individuals should have no systemic disease, should be non-smokers of cigarette or tobacco products, not in a pregnancy, have not used any antibiotics or medications with an impact on the immune system within last 6 months, have GR classified as Miller class I or class II, have GR depth of ≥2mm , have no decay or restoration on the vital teeth which will be operated, have no operation history with regard to GRs for related tooth area. The materials and methods of this study were approved by the Non-Drug Clinical Researches Ethics Committee of Yüzüncü Yıl University (B.30.2.YYU.0.01.00.00/32).

Study Groups:

In SCTG group 17 of GRs defects and in SCTG+EMD group 18 GRs defects were treated. While GRs in SCTG group was treated by SCTG and CPF combination therapy, EMD (Emdogain, Straumann, Basel, Switzerland) was additionally used in GR treatments of SCTG+EMD group. Patients were randomized by complete randomization method (SPSS 15; SPSS Inc., Chicago, IL, USA) to assign them into groups.

Pre-surgical Procedure:

Patients were informed about the potential causes of GRs. Causative habits of GR have been eliminated. Baseline periodontal treatments of the patients were performed. Plaque index (PI) , gingival index (GI) , probing pocket depth (PPD) (mm), clinical attachment level (CAL) (mm) were recorded before periodontal treatment. We prepared patients with total PI scores less than 15% for the surgical procedure (O'Leary et al 1972). Pre-treatment 3D soft tissue images were taken by CEREC Omnicam (Sirona Dental Systems GmbH, Bensheim, Germany) from intra-oral region. Recipient zone was prepared using the Langer method. SCTG was extracted ipsilaterally with the operation site from the palatal region between distal of canine and mesial of 1st molar tooth. Incision was performed in parallel with free gingival margin using Harris graft knife (Harris Double Blade Graft Knife, H & H Company, Ontario, CA, USA). Harvested graft was implanted to recipient zone so that its periosteal side faces with root surface and overhangs defect borders by 1mm. In order to remove the smear layer on the root surface of the teeth in SCTG+EMD group, 24% EDTA (Prefgel, Straumann, Basel, Switzerland) was applied for two minutes onto the root surface and operation site was washed with normal saline in order to remove any residual EDTA. EMD was applied to entire root surface compatible with manufacturer's instructions .

Post-surgical Procedure:

3D images and clinical parameter values were recorded during follow-up examinations at the 1st and the 6th month after the periodontal surgery. 3D images of soft tissue were taken intraorally with CEREC Omnicam® device at the commencement of treatment as well as at the post-operative 1st and 6th months . The measurements were recorded as in rst.img format which is a file extension of CEREC system®. The operation site was cut out from the image which was recorded at the 1st and at the 6th month. Images of each patient which were taken in three different time points were overlapped on Mimics 10 software. GGV and GGSA measurements were made on the overlapped images. the GGV and GGSA were calculated the difference in tissue as obtained after overlapping the 3D images by the software. Changes at the 1st and the 6th month after treatment were calculated with respect to pre-treatment images .

ELIGIBILITY:
Inclusion Criteria:

* individuals should have no systemic disease
* non-smokers of cigarette or tobacco products
* not in a pregnancy,
* have not used any antibiotics or medications with an impact on the immune system within last 6 months,
* have GR classified as Miller class I or class II
* have GR depth of ≥2mm ,
* have no decay or restoration on the vital teeth which will be operated
* have no operation history with regard to GRs for related tooth area.

Exclusion Criteria:

* pregnancy
* smoking
* Miller class III and IV gingival recession
* antibiotic use

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
GGV | 6 months
  Gingival gain volume: measured by software on images (mm3)
GGSA | 6 months
  Gingival gain of surface area: measured by software on images (mm2
GRH | 6 months
  gingival recession height: the distance between cementoenamel junction to gingival margin (mm)
GRW | 6 months
  gingival recession width: the distance between mesial and distal gingival margins (mm)

IPD SHARING:
Plan to Share IPD: Undecided